CLINICAL TRIAL: NCT01949077
Title: Evaluation of Serum Chemokines for Patients Undergoing Treatment With Boceprevir.
Status: Withdrawn | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-2124
Record Dates: First submitted 2013-09-10; First posted 2013-09-24 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C
Keywords: Hepatitis; Hepatitis C; Observational study; Biomarkers of treatment response
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum and tissue collected through the UNC Liver Center serum and tissue bank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sustained virological response: Patients who achieve sustained virological response (SVR) are defined as undetectable HCV RNA in serum obtained 12 weeks or beyond the end of antiviral therapy.
- Non-responders: Non-responders are defined as patients who have not achieved virological milestones during therapy or who have relapsed with detectable HCV RNA in serum after cessation of treatment.

SUMMARY:
The purpose of the study is to determine differences in levels of serum chemokines from patients undergoing treatment with Boceprevir. The aim is to determine if non-responders have significantly different levels of chemokines than responders.

DETAILED DESCRIPTION:
Patients undergoing standard of care at the UNC Liver Center are consented for collection of an additional serum sample under the UNC Liver Center serum and tissue bank study. These samples will be used to analyze differences in serum chemokines across responders and non-responders.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 or older) treated with an antiviral Hepatitis C treatment regimen that includes Boceprevir.

Exclusion Criteria:

* Inability to provide informed consent for a serum sample enrolled in the University of North Carolina Liver Center serum bank.
* No pre and post serum sample available within 6 months of the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult patients: Aged 18 and older with chronic HCV treated with triple therapy (including Boceprevir).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Level (ng/mL) of serum chemokines. | Baseline: <=6 months prior to start of treatment and Post-treatment: <=6-months after the last dose
  Compare levels of serum chemokines across Boceprevir responders (SVR) and non-responders for both Baseline (<=6-months pre-treatment) and Post-treatment (<=6-months post-treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Fried, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Liver Center, Chapel Hill, North Carolina, United States